CLINICAL TRIAL: NCT05628688
Title: A Non-randomized, Open-Label Study to Evaluate the Safety and Effectiveness of Insight® Pro Device for Evaluating Lymphatic and Venous Disorders (VOLGA)
Acronym: VOLGA
Status: Completed | Type: Observational
Sponsor: Koya Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: KCT 011 (VOLGA)
Record Dates: First submitted 2022-11-09; First posted 2022-11-29 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Lymphedema; Chronic Venous Insufficiency; Edema; Venous Insufficiency of Leg
MeSH Terms: conditions — Lymphedema; Edema | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Test group: Up to 50 subjects will be enrolled with unilateral or bilateral edema in the upper or lower extremity.
  Interventions: Diagnostic Test: Insight Pro Device for Diagnosis
- Control group: Up to 50 patients will be enrolled from a healthy volunteer group as a control, with no edema.
  Interventions: Diagnostic Test: Insight Pro Device for Diagnosis

INTERVENTIONS:
Diagnostic Test: Insight Pro Device for Diagnosis — Insight Pro Device for Diagnosis of Lymphatic and Venous Disorders

SUMMARY:
To demonstrate that the Insight Pro Device is safe and effective for use in detecting lymphatic and venous disorders.

DETAILED DESCRIPTION:
6. Clinical Hypotheses

1. The Insight Pro device can detect a difference in extracellular fluid volume through bioimpedance and dielectric constant measurement.
2. The Insight Pro device can detect a difference in skin hardness or fibrositis through a durometer measurement.
3. The Insight Pro device is safe for use as assessed by adverse events.

ELIGIBILITY:
Inclusion Criteria:

Test group -

* Males and females ≥ 18 years of age
* Willing to sign the informed consent and deemed capable of following the study protocol
* Subjects must have primary or secondary unilateral or bilateral upper or lower extremity edema
* At the time of initial evaluation, individuals must be at least 3 months post-surgery, chemotherapy and/or radiation treatment for cancer if applicable

Control group -

* Males and females ≥ 18 years of age
* Willing to sign the informed consent and deemed capable of following the study protocol
* Subjects must not have primary or secondary edema and self-describe general healthy

Exclusion Criteria:

* ● Inability or unwillingness to participate in all aspects of the study protocol and/or failure to provide informed consent

  * Patients with exam results that would prevent safe and effective use of the study device (cellulitis, open-wounds, healing-wounds, etc.)
  * Diagnosis of active or recurrent cancer (< 3 months since completion of chemotherapy, radiation therapy, or primary surgery for the cancer)
  * Patients with cardiac arrhythmia with pacemakers or other implanted electronic equipment
  * Patients must not have implanted metal hardware in the limbs
  * Patients undergoing external defibrillation
  * Diagnosis of Acute infection (in the last four weeks)
  * Diagnosis of acute thrombophlebitis (in last 2 months)
  * Diagnosis of pulmonary embolism or deep vein thrombosis within the previous 2 months
  * Diagnosis of congestive heart failure (uncontrolled)
  * Diagnosis of chronic kidney disease with acute renal failure
  * Women who are pregnant, planning a pregnancy or nursing at study entry
  * Participation in any clinical trial of an investigational substance or device during the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: (Test Group) - Up to 50 subjects will be enrolled with unilateral or bilateral edema in the upper or lower extremity.
  (Control Group) Up to 50 patients will be enrolled from a healthy volunteer group as a control, with no edema.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
Edema Volume | Acute - At day 0
  Edema Volume detection by difference in extracellular fluid volume through bioimpedance and dielectric constant measurement.
Fibrosis | Acute - At day 0
  Durometer detection or Skin hardness (fibrosis) difference through a durometer measurement.

SECONDARY OUTCOMES:
Safety/AEs | Acute - At day 0
  Safety during use (via adverse event reporting)
LymVAS | Acute - At day 0
  Correlation with quality-of-life objective parameters using a lymphedema visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- Koya Medical, Inc., Oakland, California, United States

IPD SHARING:
Plan to Share IPD: Undecided